CLINICAL TRIAL: NCT00610961
Title: The Induction Agent Effect on BK Viremia in Renal and Pancreas Transplant Patients
Brief Title: Induction Related BK Viremia in Renal Transplant Patients
Acronym: BK
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 20071016
Record Dates: First submitted 2008-01-24; First posted 2008-02-08 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Disease Due to BK Polyomavirus; Transplantation Infection; Disorder Related to Transplantation
Keywords: BK Polyomavirus; Transplantation, Kidney; Transplantation, Pancreas

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Basiliximab (Simulect) Induction: Prospective group: patients are scheduled to receive a kidney transplant; and will receive Simulect®, Myfortic® and Prograf® with or without steroids according to routine care (Standard of Care).
- Thymoglobulin Induction: Retrospective (historical or control) group: patients have already received a kidney transplant and were treated with Thymoglobulin®, Myfortic®, and Prograf® with or without steroids. This treatment was Standard of Care at a time of transplant.

SUMMARY:
The increase immunosuppression in our transplant population has led to an unacceptable rate of patients at risk for BK virus nephropathy. Reducing induction immunosuppression by switching from Thymoglobulin to Simulect will reduce the incidence of serum positivity for BK by PCR.

DETAILED DESCRIPTION:
Our standard of care has been changed from Thymoglobulin to Simulect and now patients were enrolled in this observational trial to gather data on their outcomes related to BK viremia and rejection rates. Two groups of patients were compared.

Retrospective (historical or control) group of subjects: patients who had received a kidney transplant and were inducted with Thymoglobulin prior to study initiation.

Prospective group of subjects: patients who is scheduled to receive kidney transplant and will be inducted with Simulect (Basiliximab).

Inductions in both groups was/is Standard of Care at a time of treatment.

ELIGIBILITY:
Inclusion Criteria:

* De novo transplant
* Aged 18-75

Exclusion Criteria:

* Serious medical condition which, in the opinion of the Principal Investigator, might interfere with the subject's ability to successfully complete the protocol.
* Any medical condition which, in the opinion of the Principal Investigator, might compromise the safety of the subject in participating in the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: de novo renal or renal/pancrease transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
BK Virus Viremia titer, >400 copies by Polymerase Chain Reaction (PCR) | One year
  BKVV (BK Visus Viremia) titer is measured by PCR at 1, 3,6,9 and 12 month time points.

SECONDARY OUTCOMES:
Incidence of Acute Rejection of Transplanted Kidney | One year

CONTACTS AND LOCATIONS:
Overall Officials: Herwig-Ulf Meier-Kriesche, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States